CLINICAL TRIAL: NCT01803607
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Odanacatib (MK-0822) on Bone Mineral Density (BMD) and Overall Safety in the Treatment of Osteoporosis in Postmenopausal Women Previously Treated With an Oral Bisphosphonate
Brief Title: Efficacy and Safety of Odanacatib in Postmenopausal Women Previously Treated With Oral Bisphosphonate (MK-0822-076)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely due to low enrollment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-076
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Odanacatib 50 mg (Experimental): Participants will receive odanacatib 50 mg once weekly for 24 months. Additionally, all participants will receive weekly supplementation with 5600 international units (IU) of Vitamin D3 and, if required, will be provided with an open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium.
  Interventions: Drug: odanacatib
- Placebo (Placebo Comparator): Participants will receive dose-matched placebo to odanacatib once weekly for 24 months. Additionally, all participants will receive weekly supplementation with 5600 IU Vitamin D3 and, if required, will be provided with an open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium.
  Interventions: Other: placebo to odanacatib

INTERVENTIONS:
Drug: odanacatib — odanacatib 50 mg oral tablet
  Other Names: MK-0822
  Arms: Odanacatib 50 mg
Other: placebo to odanacatib — dose-matched placebo to odanacatib, oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess to what extent sequential treatment with odanacatib results in incremental gains in bone mineral density (BMD) over time in female participants who have received at least 3 years of bisphosphonate therapy. It was hypothesized that odanacatib treatment would increase femoral neck BMD relative to placebo after 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for ≥5 years (defined as no menses for at least 5 years or at least 5 years post bilateral oophorectomy).
* Prior or current treatment with oral bisphosphonate therapy (i.e., alendronate, risedronate, ibandronate) for postmenopausal osteoporosis for ≥3 years.
* BMD T-score at any hip site (femoral neck, trochanter, or total hip) ≤-2.5 and >-3.5 as assessed by dual-energy X-ray absorptiometry (DXA) without a history of a prior fragility fracture. For participants with a history of a prior fragility fracture (except hip fracture), BMD T-score can be ≤-1.5 and >-3.5 at any hip site.
* Serum 25-hydroxyvitamin D level of ≥20 and ≤60 ng/mL within 90 days of the time of randomization.

Exclusion Criteria:

* Evidence of a metabolic bone disorder other than osteopenia or osteoporosis
* History or current evidence of hip fracture.
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Active parathyroid disease. Participant with a documented history of parathyroid disease can be considered for inclusion if she has normal parathyroid hormone (PTH) at screening.
* History of thyroid disease not adequately controlled by medication.
* Current treatment with anti-seizure medication, with indices of calcium metabolism not within normal limits.
* Prior treatment with strontium-containing products; intravenous bisphosphonates; cathepsin K inhibitors; RANK ligand inhibitors; fluoride treatment at a dose greater than 1 mg/day for more than 2 weeks.
* Use of following medications within the 6 months prior to the screening visit: activated vitamin D; estrogen, with or without progestin, at a dose high enough to have systemic effects; raloxifene or other selective estrogen receptor modulator (SERM), tibolone or any aromatase inhibitor; sub-cutaneous calcitonin (Note: use of intranasal calcitonin is allowed at any time); anabolic steroid; PTH (1-34 or 1-84); growth hormone; systemic glucocorticoids (≥5 mg/day of prednisone or equivalent) for more than 2 weeks; cyclosporine for more than 2 weeks.
* Concurrent use of cancer chemotherapy or heparin; protease inhibitors for human immunodeficiency virus (HIV) treatment; and vitamin A (excluding beta carotene) >10,000 IU daily, unless willing to discontinue this dose during the study.
* Current treatment with cytochrome P450 3A4 (CYP3A4) inducers or treatment with CYP3A4 inducer within 4 weeks of screening.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2014-11-11 (Actual); Study Completion 2014-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal female participants ≥60 years of age with low bone mineral density (BMD) and who had been treated with an oral bisphosphonate for at least 3 years were recruited at 81 sites in the United States.
Pre-assignment Details: The Sponsor made a business decision to terminate the trial early due to poor enrollment; the decision was not related to any findings regarding the efficacy or safety profile of odanacatib.
Groups:
- Odanacatib 50 mg: Participants received odanacatib 50 mg OW for 24 months. In addition, participants received Vitamin D 5600 IU as well as open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium.
- Placebo: Participants received dose-matched placebo to odanacatib OW for 24 months. In addition, participants received Vitamin D 5600 IU as well as open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium.
Period: Overall Study
Arm/Group | Odanacatib 50 mg | Placebo
Started | 68 | 67
Completed | 0 | 0
Not Completed | 68 | 67
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Study terminated by sponsor | 54 | 56
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Odanacatib 50 mg | Placebo | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (7.9) | 70.7 (7.6) | 70.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 135
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 12 in Femoral BMD
Description: Dual-energy X-ray absorptiometry (DXA) was used to determine the change from baseline in femoral neck BMD at Month 12.
Time Frame: Baseline and Month 12
Population: The Full Analysis set (FAS) includes all randomized participants who took at least one dose of study medication and had the relevant baseline and follow-up measurements.
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 24 | 20
Percent Change from Baseline | 0.70 (1.00) | -0.20 (1.17)

2. Secondary Outcome: Percent Change From Baseline to Month 24 in Femoral Neck BMD: Within-Group Comparison of Odanacatib
Description: DXA was used to determine the within-group change from baseline in femoral neck BMD at Month 24.
Time Frame: Baseline and Month 24
Population: The trial was terminated prematurely, thus this analysis was not conducted.
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Baseline to Month 12 in Trochanter, Total Hip, and Lumbar Spine BMD
Description: DXA was used to determine the change from baseline in trochanter, total hip, and lumbar spine BMD at Month 12.
Time Frame: Baseline and Month 12
Population: The FAS includes all randomized participants who took at least one dose of study medication and had the relevant baseline and follow-up measurements
Measure: Mean (Standard Error); unit: Percentage Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 24 | 20
Percentage Change from Baseline
  Trochanter | 1.85 (1.14) | -1.66 (1.13)
  Total Hip | -0.09 (0.63) | -1.67 (0.51)
  Lumbar Spine | 2.10 (0.99) | -1.52 (0.86)

4. Secondary Outcome: Change From Baseline in Serum C-telopeptides of Type 1 Collagen (s-CTx)
Description: s-CTx is a biochemical marker of bone resorption. At baseline and Month 12, s-CTx was measured and expressed in ng/mL and results are expressed as percentage change from baseline.
Time Frame: Baseline and Month 12
Population: The Per Protocol (PP) population includes all participants who received 1 dose of study drug, had the necessary baseline and post-baseline data, and did not have any protocol violations that may substantially impact results.
Measure: Geometric Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 18 | 23
Percent Change from Baseline | 15.37 (20.24) | 44.10 (10.19)

5. Secondary Outcome: Change From Baseline in Urine C-telopeptides of Type I Collagen (u-CTx)
Description: u-CTx is a biochemical marker of bone resorption. At baseline and Month 12, u-CTx was measured and expressed in ug/mL and results are expressed as percentage change from baseline.
Time Frame: Baseline and Month 12
Population: The PP population includes all participants who received 1 dose of study drug, had the necessary baseline and post-baseline data, and did not have any protocol violations that may substantially impact results.
Measure: Geometric Mean (Standard Error); unit: Percentage Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 17 | 20
Percentage Change from Baseline | -82.39 (22.46) | 63.21 (23.08)

6. Secondary Outcome: Change From Baseline in Urine N-telopeptides of Type 1 Collagen Corrected for Creatinine (u-NTx/Cr)
Description: The u-NTx/Cr ratio is a biochemical marker of bone resorption. u-NTx/Cr was measured at baseline and Month 12 and expressed in nM:mM and results are expressed as percentage change from baseline.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Geometric Mean (Standard Error); unit: Percentage Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 17 | 22
Percentage Change from Baseline | -29.78 (13.46) | 37.73 (10.46)

7. Secondary Outcome: Change From Baseline in Serum Bone Specific Alkaline Phosphatase (s-BSAP)
Description: s-BSAP is a biochemical marker of bone resorption. s-BSAP was measured and expressed in ng/mL at Baseline and Month 12, and results are shown as percentage change from baseline.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Geometric Mean (Standard Error); unit: Percentage Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 18 | 23
Percentage Change from Baseline | 22.32 (7.91) | 17.19 (4.09)

8. Secondary Outcome: Change From Baseline in Serum N-terminal Propeptide of Type 1 Collagen (s-P1NP)
Description: s-P1NP is a biochemical marker of bone resorption. s-P1NP was measured and expressed as ng/mL at Baseline and Month 12, and results are expressed as percentage change from baseline.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Geometric Mean (Standard Error); unit: Percentage Change from Baseline
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 18 | 23
Percentage Change from Baseline | 53.65 (16.91) | 56.15 (8.80)

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: An AE is any unfavorable and unintended change in the structure (signs), function (symptoms), or chemistry (laboratory data) of the body temporally associated with any use of a Sponsor product, whether or not considered related to the use of the product.
Groups:
- ODN 50 mg OW: Participants received odanacatib 50 mg OW for 24 months. In addition, participants received Vitamin D 5600 IU as well as open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium.
- Placebo OW: Participants received dose-matched placebo to odanacatib OW for 24 months. In addition, participants received Vitamin D 5600 IU as well as open-label daily calcium supplement of 500 mg (sourced locally as calcium carbonate or calcium citrate) to ensure a total daily intake (from both dietary and supplemental sources) of approximately 1200 mg of elemental calcium. One participant who was randomized to odanacatib 50 mg OW received placebo during the entire treatment period and was therefore included in the Placebo OW group for safety analyses.
Arm/Group | ODN 50 mg OW | Placebo OW
Serious Adverse Events (participants affected / at risk) | 6/67 | 4/68
Other Adverse Events (participants affected / at risk) | 15/67 | 9/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODN 50 mg OW (N=67) | Placebo OW (N=68)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODN 50 mg OW (N=67) | Placebo OW (N=68)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (7) | 3 (5)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.